CLINICAL TRIAL: NCT03627026
Title: Evaluation of Sphingolipids as Predictive Biomarkers of Immune Checkpoint Inhibitor Response in Melanoma Patients
Acronym: IMMUSPHINX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18 CUTA 05
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Melanoma
Keywords: Melanoma; Sphingolipids; Immune checkpoints; Tumor-infiltrating lymphocytes; Immunosuppressive cytokines; Circulating leukocytes
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with immune checkpoint inhibitor (Other)
  Interventions: Other: Blood samples will be collected at different time points:

INTERVENTIONS:
Other: Blood samples will be collected at different time points: — * Baseline
  * Week 6 Day 1
  * Week 12 Day 1
  If feasible, an optional tumor biopsy specimen will be collected during baseline visit for a maximum of 30 patients included in IUCT-O center.

SUMMARY:
This trial is a translational proof-of-concept, open-label, prospective cohort study of 60 patients aiming to identify the clinical markers and/or biomarkers associated with therapeutic response to immune checkpoints inhibitors, in patients with advanced melanoma.

The study will be conducted on a population of patients treated with anti-PD-1 alone (nivolumab or pembrolizumab) or in combination (nivolumab + ipilimumab) in the context of routine care.

For each included patient, blood samples will be collected at different time points.

If feasible, an optional tumor biopsy specimen will be collected during baseline visit.

All included patients will be followed-up for tumor response and toxicity until Week 12.

After Week 12, survival data (tumor status and/or survival status) will be collected every 3 months until a maximum duration of 1 year from the first study dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of study entry.
2. Patient with histologically-proven metastatic and/or unresectable melanoma (stage IIIc-IV, M1a-c as per AJCC 8th edition), including mucosal melanoma, without intracranial active disease.
3. Patient for which a treatment with immune checkpoint inhibitor (nivolumab alone, pembrolizumab alone, nivolumab plus ipilimumab) has been decided.
4. Subjects are included regardless of BRAFV600 mutation status. BRAFV600 mutation status must be documented.
5. Patient must be naïve to immune checkpoint inhibitor treatment for locally advanced and/or metastatic disease (i.e., no prior treatment with ICI and current treatment with ICI not yet started).
6. ECOG Performance status 0-2.
7. Life expectancy of at least 3 months.
8. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol.
9. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Patient pregnant, or breast-feeding.
2. Uveal melanoma.
3. Any condition contraindicated with sampling procedures required by the protocol.
4. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
5. Any current severe or uncontrolled disease, including, but not limited to ongoing or active infection.
6. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the discriminant capacity to predict progression at 12 weeks evaluated using RECIST V1.1 criteria. | 12 weeks per patient

SECONDARY OUTCOMES:
Objective response (i.e. complete or partial response) will be defined using RECIST V1.1 criteria at week 12. | 12 weeks per patient
Response duration is defined as the time from objective response until progression according to investigator judgment, or death. | 12 months per patient
Progression Free Survival is defined as the time from inclusion until progression according to investigator judgment, or death, whichever occurs first. | 12 months per patient

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Nantes, Nantes
  - Institut Universitaire Du Cancer de Toulouse - Oncopole, Toulouse